CLINICAL TRIAL: NCT02019108
Title: Effects of Toe-out Gait Modification on Clinical and Biomechanical Measures in People With Knee Osteoarthritis
Brief Title: Gait Modification Treatment for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Melbourne (Other); Arthritis Research Centre of Canada (Other)
Responsible Party: Principal Investigator, Michael Hunt, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-02688; SOG-13-024 (Other Grant/Funding Number: The Arthritis Society (Canada))
Record Dates: First submitted 2013-12-05; First posted 2013-12-24 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee; walking; toeout; gait modification
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait Modification Group (Experimental): Participants will complete 4 months of a home-based progressive walking program with toe-out gait modification aimed at improving physical activity level. This group will perform continuous treadmill walking during regular sessions with a study therapist and will be instructed to perform a toe-out gait, with the aid of a mirror during walking. Focus will also be on increasing the time and distance of walking. These goals will be emphasized for the home-based portion of the intervention as well.
  Interventions: Other: Progressive walking program with toe-out gait modification
- Walking Only Group (Active Comparator): Participants will complete 4 months of a home-based progressive walking program aimed at improving physical activity level. This group will perform continuous treadmill walking during regular sessions with the study therapist with focus on increasing the time and distance of walking. This goal will be emphasized for the home-based portion of the intervention as well.
  Interventions: Other: Progressive walking program

INTERVENTIONS:
Other: Progressive walking program with toe-out gait modification — Participants in this study group will perform continuous treadmill walking for a minimum of 30 minutes at each session, but the emphasis will be to increase toe-out angle by 10 degrees over that exhibited at baseline. A mirror will be provided for biofeedback and participants will be instructed on its use for achieving the target toe-out angle. Increased walking time and distance will be encouraged the same as for the control group.
  Arms: Gait Modification Group
Other: Progressive walking program — At each scheduled visit, participants will perform treadmill walking for a minimum of 30 minutes depending on the individual's baseline activity level and the stage of the intervention. Emphasis will be solely on increasing walking time and distance to achieve the target of a 40% increase in daily activity.
  Arms: Walking Only Group

SUMMARY:
Knee osteoarthritis (OA) is a costly health condition affecting more than 10% of Canadian adults. Excessive and unbalanced loads passing through the knee joint have been implicated in the progression of OA. Typical conservative treatment of OA has focused on increasing daily activity, without consideration for the underlying joint loading. This study aims to compare a 4-month walking program that aims to increase the angle of the foot (toe-out angle) during walking - a measure shown to reduce joint loading and OA disease progression - while increasing walking time/distance, with a standard walking program that aims to increase walking time/distance. It is predicted that the walking program focusing on increasing toe-out will provide greater reductions in self-reported knee pain and a greater reduction in unfavorable knee joint loading.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 years and older
* radiographically confirmed medial compartment tibia-femoral knee osteoarthritis
* available for weekly training sessions in the Vancouver British Columbia Canada region
* able to safely perform treadmill walking under therapist supervision

Exclusion Criteria:

* articular cartilage degradation in the lateral tibiofemoral compartment greater than the medial
* inflammatory arthritic condition
* history of knee replacement or arthroscopic knee surgery
* recent use of corticosteroids (oral or via injection)
* inability to ambulate without a gait aid
* non-English speaking
* planning to commence a new treatment approach within the next 4 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Hunt, PT, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- Motion Analysis and Biofeedback Laboratory, The University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Hunt MA, Charlton JM, Krowchuk NM, Tse CTF, Hatfield GL. Clinical and biomechanical changes following a 4-month toe-out gait modification program for people with medial knee osteoarthritis: a randomized controlled trial. Osteoarthritis Cartilage. 2018 Jul;26(7):903-911. doi: 10.1016/j.joca.2018.04.010. Epub 2018 Apr 27. PMID 29709498

RESULTS

PARTICIPANT FLOW:
Groups:
- Gait Modification Group: Participants will complete 4 months of a home-based progressive walking program with toe-out gait modification aimed at improving physical activity level. This group will perform continuous treadmill walking during regular sessions with a study therapist and will be instructed to perform a toe-out gait with the aid of a mirror during walking. Focus will also be on increasing the time and distance of walking. These goals will be emphasized for the home-based portion of the intervention as well.
  Progressive walking program with toe-out gait modification: Participants in this study group will perform continuous treadmill walking for a minimum of 30 minutes at each session, but the emphasis will be to increase toe-out angle by 10 degrees over that exhibited at baseline. A mirror will be provided for biofeedback and participants will be instructed on its use for achieving the target toe-out angle. Increased walking time and distance will be encouraged the same as for the control group.
Period: Overall Study
Arm/Group | Gait Modification Group | Walking Only Group
Started | 40 | 39
Baseline (Week 0) | 40 | 39
Follow-up (Week 17) | 38 | 36
Retention (Week 21) | 35 | 32
Completed | 35 | 32
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gait Modification Group | Walking Only Group | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (7.6) | 65.4 (9.6) | 65.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 13 | 11 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 39 | 79
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (3.5) | 27.4 (3.5) | 27.4 (3.5)
Radiographic Severity [Count of Participants; unit: Participants] — Kellgren and Lawrence grading criteria for mild (grade 2), moderate (grade 3), and severe (grade 4) radiographic osteoarthritis.
  Participants
    Mild (KL2) | 19 | 18 | 37
    Moderate (KL3) | 17 | 14 | 31
    Severe (KL4) | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Pain as Measured by Numerical Rating Scale
Description: Average pain over the previous week will be assessed using an 11-point numerical rating scale (0 = no pain; 10 = maximum pain). Higher scores mean a worse outcome. Change was calculated as the value at 17 weeks and at 21 weeks minus the value at baseline.
Time Frame: Weeks 0, 17, 21
Population: Participants lost to follow-up. Gait modification group lost 2 participants by week 17 and 3 additional participants by week 21 making a total loss of 5. Walking Only group lost 3 participants by week 17 and 4 additional participants by week 21 making a total loss of 7.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 38 | 36
units on a scale
  Change from Baseline to Week 17 | -2.1 [-2.7 to -1.5] | -1.8 [-2.4 to -1.2]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 32
  Change from Baseline to Week 21 | -2.2 [-2.8 to -1.7] | -1.5 [-2.1 to -0.9]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p = 0.495, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.1 to 0.5]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.079, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.6 to 0.1]

2. Primary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale.
Description: Lower-limb impairments will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC is a 24-item self-report questionnaire that quantifies pain (5 items), stiffness (2 items), and physical function (17 items). It is a valid, reliable, and responsive disease-specific self-report instrument and has been used in many knee OA studies. Minimum value of the WOMAC pain subscale is 0 and maximum value is 20. Higher scores mean a worse outcome.
Time Frame: Weeks 0, 17, 21
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 38 | 36
units on a scale
  Change from Baseline to Week 17 | -2.7 [-3.6 to -1.7] | -1.5 [-2.5 to -0.5]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 32
  Change from Baseline to Week 21 | -2.5 [-3.5 to -1.6] | -1.5 [-2.5 to -0.5]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p = 0.117, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.6 to 0.3]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.133, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.5 to 0.3]

3. Primary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Knee Joint Loading: First Peak Knee Adduction Moment
Description: Participants will undergo a gait analysis, where 10-15 trials of walking will be collected. Participants will walk in bare feet and at their own, self-selected speed while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and floor-mounted force platforms. A total of 5 "acceptable" (clean force platform strikes and no observable deviation in walking characteristics) will be analyzed.
Time Frame: Weeks 0, 17, 21
Population: Participants lost to follow-up. Gait modification group lost 3 participants by week 17 and 2 additional participants by week 21 making a total loss of 5. Walking Only group lost 6 participants by week 17 and 2 additional participants by week 21 making a total loss of 8.
Measure: Least Squares Mean (95% Confidence Interval); unit: %Body Weight*Height
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 37 | 33
%Body Weight*Height
  Change from Baseline to Week 17 | -0.01 [-0.13 to 0.11] | 0.13 [0.00 to 0.26]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 31
  Change from Baseline to Week 21 | -0.06 [-0.20 to 0.08] | 0.11 [-0.04 to 0.26]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p = 0.125, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Median Difference (Final Values) = -0.14, 95% CI 2-sided [-0.31 to 0.04]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.103, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.37 to 0.03]

4. Primary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Knee Joint Loading: Second Peak Knee Adduction Moment
Description: as for outcome 3
Time Frame: Weeks 0, 17, 21
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: %Body Weight*Height
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 37 | 33
%Body Weight*Height
  Change from Baseline to Week 17 | -0.24 [-0.33 to -0.15] | 0.02 [-0.08 to 0.11]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 31
  Change from Baseline to Week 21 | -0.19 [-0.33 to -0.04] | 0.01 [-0.14 to 0.16]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p < 0.001, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.39 to -0.12]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.056, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.40 to 0.01]

5. Primary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Knee Joint Loading: Knee Adduction Moment Impulse
Description: as for outcome 3
Time Frame: Weeks 0, 17, 21
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: %Body Weight*Height*seconds
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 37 | 33
%Body Weight*Height*seconds
  Change from Baseline to Week 17 | -0.04 [-0.08 to -0.01] | 0.01 [-0.02 to 0.05]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 31
  Change from Baseline to Week 21 | -0.06 [-0.10 to -0.02] | 0.00 [-0.04 to 0.05]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p = 0.031, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.11 to -0.01]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.058, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.12 to 0.00]

6. Primary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Foot Progression Angle (FPA)
Description: FPA indicates orientation of the foot with respect to the forward progression of the body. Positive values correspond to a toe-in orientation, whereas negative values correspond to a toe-out orientation. Therefore, a positive change value indicates more toe-in versus a negative change value indicates more toe-out.
Time Frame: Weeks 0, 17, 21
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 37 | 33
degrees
  Change from Baseline to Week 17 | -8.87 [-10.36 to -7.39] | 0.17 [-1.41 to 1.74]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 31
  Change from Baseline to Week 21 | -6.96 [-8.35 to -5.58] | -0.18 [-1.66 to 1.29]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p < 0.001, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -9.04, 95% CI 2-sided [-11.22 to -6.86]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p < 0.001, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -6.78, 95% CI 2-sided [-8.82 to -4.75]

7. Secondary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Self-reported Physical Function as Measured by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale.
Description: Lower-limb impairments will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC is a 24-item self-report questionnaire that quantifies pain (5 items), stiffness (2 items), and physical function (17 items). It is a valid, reliable, and responsive disease-specific self-report instrument and has been used in many knee OA studies. The WOMAC physical function subscale minimum value is 0 and maximum value is 68. Higher scores mean a worse outcome.
Time Frame: Weeks 0, 17, 21
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 38 | 36
units on a scale
  Change from Baseline to Week 17 | -11.4 [-14.6 to -8.3] | -7.7 [-10.9 to -4.5]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 32
  Change from Baseline to Week 21 | -9.4 [-12.4 to -6.3] | -6.6 [-9.8 to -3.4]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p = 0.111, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-8.3 to 0.9]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.232, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-7.3 to 1.8]

8. Secondary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Objective Physical Function as Measured by Timed Stair Climb.
Description: Participants were instructed to ascend 12 stairs "as quickly as possible", and the fastest time from two attempts was recorded.
Time Frame: Weeks 0, 17, 21
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 37 | 33
seconds
  Change from Baseline to Week 17 | -0.16 [-0.55 to 0.24] | -0.37 [-0.78 to 0.05]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 31
  Change from Baseline to Week 21 | -0.44 [-0.89 to 0.01] | -0.33 [-0.80 to 0.14]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p = 0.462, ANCOVA — a priori threshold for significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.36 to 0.78]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.737, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.76 to 0.54]

9. Secondary Outcome: Change From Baseline to Week 17 and From Baseline to Week 21 in Knee Joint Loading: Knee Flexion Moment
Description: as for outcome 3
Time Frame: Weeks 0, 17, 21
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: %Body Weight*Height
Arm/Group | Gait Modification Group | Walking Only Group
Number analyzed (Participants) | 37 | 33
%Body Weight*Height
  Change from Baseline to Week 17 | 0.06 [-0.26 to 0.38] | 0.09 [-0.24 to 0.43]
  Change from Baseline to Week 21: number analyzed (Participants) | 35 | 31
  Change from Baseline to Week 21 | 0.31 [-0.01 to 0.62] | 0.28 [-0.06 to 0.61]
Statistical Analysis 1: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 17 weeks; Test type: Superiority; p = 0.876, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.50 to 0.43]
Statistical Analysis 2: Comparison: Gait Modification Group vs Walking Only Group; This is the comparison between Gait Modification Group and Walking Only Group at 21 weeks; Test type: Superiority; p = 0.897, ANCOVA — a priori threshold for statistical significance <0.05; Controlling for baseline values and walking speed; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.43 to 0.49]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during weeks 1 - 16 by diary entry and at each visit (Weeks 1, 2, 4, 6, 8, 10, 12 and 15) with the study trainer.
Description: Adverse event data collected by participant self-report.
Arm/Group | Gait Modification Group | Walking Only Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 8/40 | 4/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gait Modification Group (N=40) | Walking Only Group (N=39)
Hip Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Big Toe Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Posterior Thigh Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT02019108/Prot_SAP_000.pdf